CLINICAL TRIAL: NCT03571906
Title: Tele - Cardiac Rehabilitation - Providing Pre-habilitation to Stable Patients With Valvular Heart Disease Awaiting Surgery
Brief Title: Pre-habilitation of Patients Scheduled for Cardiac Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Prof. Klempfner, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4517-17-SMC
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Valvular Heart Disease
Keywords: Rehabilitation
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-rehab intervention (Experimental): Subjects in the prehab arm will receive an exercise prescription and execution will be assessed and periodically adjusted in accordance to data received from the wearable device. Intensity and type of exercise will be moderate and will comply with exercise recommendations provided by ESC guidelines. A dedicated application will be installed on the mobile phone for patients in the research group and they will receive a smart sports watch.
  Periodic encouragements and consultations will be provided by exercise trainer, physiologist and nurse from the cardiac rehabilitation center. A physician will be available for consultations.
  In addition to monitored physical activity, patients will receive nutritional and psychological counseling. This is part of a multi-professional rehabilitation program accepted by the rehabilitation center.
  Interventions: Behavioral: Tele - Cardiac Pre-Rehabilitation
- pre-operative usual care arm (No Intervention): The control group will receive recommendations for a healthy and active lifestyle and physician follow-up
  All subjects will undergo a stress test at baseline (post enrollment), and again prior to cardiac surgery.

INTERVENTIONS:
Behavioral: Tele - Cardiac Pre-Rehabilitation — We intend to enroll 50 stable subjects with valvular heart disease scheduled for surgical intervention. Following a comprehensive clinical and physiological evaluation subjects will be randomized (1:1) to a Prehab arm (PHB) vs. usual care (UC). Subjects in the prehab arm will receive a hybrid institution and home-based exercise prescription, nutritional and psychological intervention and periodic calls. Adherence will be assessed and encouraged by smartwatch and matching smartphone software. In the usual care arm subjects will receive general recommendations following the baseline stress test performed by both groups (prehab is not standard of care or guideline based). Another stress test will be performed days prior to valve surgery Adherence to the rehab program will be assessed and a structured motivational program and follow-up will be provided in order to maximize goal completion.
  Other Names: Pre-rehab program
  Arms: Pre-rehab intervention

SUMMARY:
Cardiac rehabilitation (CR) is an integral part of cardiovascular disease management incorporating aspects of scientifically constructed appropriate physical exercise. CR has been repeatedly shown to significantly improve functional capacity, depression and wellbeing, even following short term interventions. Functional capacity is closely related to frailty, a key prognostic factor in subjects undergoing cardiac surgery. We intend to enroll 50 stable subjects with valvular heart disease scheduled for surgical intervention. Our hypothesis is that the Prehab group will improve their functional capacity to a greater degree than the usual care group, possibly associated with better clinical outcomes.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is an integral part of cardiovascular disease management incorporating aspects of scientifically constructed appropriate physical exercise, dietary intervention, secondary prevention by pharmacotherapy, and psychological intervention. CR has been repeatedly shown to significantly improve functional capacity, depression and wellbeing, even following short term interventions (6-8 weeks in accordance with the date of surgery determined for the patient.) Functional capacity is closely related to frailty, a key prognostic factor in subjects undergoing cardiac surgery. Small studies have demonstrated possible benefits of pre-habilitation - a multidisciplinary intervention aimed at improving frailty in the weeks prior to surgery.

We intend to enroll 50 stable subjects with valvular heart disease scheduled for surgical intervention. Following a comprehensive clinical and physiological evaluation subjects will be randomized (1:1) to a Prehab arm (PHB) vs. usual care (UC). Subjects in the prehab arm will receive a hybrid institution and home-based exercise prescription, nutritional and psychological intervention and periodic calls. Adherence will be assessed and encouraged by smartwatch and matching smartphone software. In the usual care arm subjects will receive general recommendations following the baseline stress test performed by both groups (prehab is not standard of care or guideline based). Another stress test will be performed days prior to valve surgery.

Our hypothesis is that the Prehab group will improve their functional capacity to a greater degree than the usual care group, possibly associated with better clinical outcomes.

The primary efficacy outcome will be exercise capacity (assessed by symptom limited stress test - estimated METS) change from baseline (enrollment) to pre-surgery evaluation visit (pre-op test).

Secondary measures:

Compare the 2 study arms in regard to:

1. Length of ICU and hospital stay
2. Perioperative adverse events
3. 30-day mortality or re-hospitalization
4. QOL and satisfaction

Patient / Group numbers: A total of 50 patients with established valvular disease will be enrolled to PHB or UC after eligibility verification by cardiothoracic surgeon

Hardware: Standard off the shelf Polar sports watch (M430) with matching smartphone software. No clinical or identifiable data will be inputted into these systems (coded subject ID only).

Clinical data and the entire program will be managed through the hospital electronic medical record (EMR). All clinical decisions \ recommendations and events will be recorded in the EMR.

Intervention: Patients will be randomized to pre-operative usual care or rehabilitation program comprising of on-site (Sheba MC) and off-site training sessions. Adherence to the rehab program will be assessed and a structured motivational program and follow-up will be provided in order to maximize goal completion.

Following the standard rehabilitation intake process (stress test, physician visit, nurse intake), the subjects in the prehab arm will receive physiologic consultation based on clinical stress tests and clinical data passed from the physician. Subjects in the prehab arm will receive an exercise prescription and execution will be assessed and periodically adjusted in accordance to data received from the wearable device. Intensity and type of exercise will be moderate and will comply with exercise recommendations provided by ESC guidelines. A dedicated application will be installed on the mobile phone for patients in the research group and they will receive a smart sports watch.

Periodic encouragements and consultations will be provided by exercise trainer, physiologist and nurse from the cardiac rehabilitation center. A physician will be available for consultations.

In addition to monitored physical activity, patients will receive nutritional and psychological counseling. This is part of a multi-professional rehabilitation program accepted by the rehabilitation center.

The control group will receive recommendations for a healthy and active lifestyle and physician follow-up

All subjects will undergo a stress test at baseline post enrollment and again prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet all the following inclusion criteria during the initial screening visit of the study (visit 1):

* Valvular heart disease and planed surgery within the next 4-12 weeks
* Age ≥ 21
* Smartphone with internet connection
* Willing and able to comply with study protocol and
* Able to follow the personalized exercise prescription, utilize Polar watch and upload exercise data per protocol

Exclusion Criteria:

Eligible patients must meet none of the following exclusion criteria:

* Advanced Heart failure (NYHA >3) or unresolved significant arrhythmia (i.e. symptomatic atrial fibrillation)
* Significant neurological or cognitive impairment
* Women of child-bearing potential
* Symptomatic hypotension, orthostatic hypotension or repeated blood pressure systolic value <100 mmHg without symptoms
* ACS or percutaneous coronary intervention (PCI) within 30 days prior to screening, or having undergone CABG surgery within 30 days prior to screening
* Inability to perform a stress test due to physical limitations
* Severe angina pectoris as defined by CCS >2
* Pulmonary disease of severity greater than mild (COPD, Asthma, ILD, CTD with lung involvement) or chronic pulmonary thromboembolic disease (CTED)
* Severe orthopedic limitations not permitting exercise
* Active myocarditis, constrictive pericarditis, restrictive or hypertrophic cardiomyopathy
* Significant anemia (Hb < 9 mg/dl)
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
* Any illness which reduces life expectancy to less than 1 year from screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in METS | 6-8 weeks
  Exercise capacity change as assessed by stress test

SECONDARY OUTCOMES:
Hospitalisation duration | 2 weeks peri-op
  Total hospital stay
ICU duration | 2 weeks peri-op
  Time spent in the post operation ICU unit
Peri operative complication | 2 weeks peri-op
  Occurrence of adverse events including pneumonia, bleeding, atrial fibrillation, Other infections